CLINICAL TRIAL: NCT02883439
Title: Open Label Two -Treatment Half Side Comparative Study to Analyse Difference in Bioavailability Between MP29-02 and Fluticasoen Propionate
Brief Title: Study to Analyse Difference in Bioavailability Between MP29-02 and Fluticasone Propionate
Acronym: BIODYMF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no available patients
Sponsor: University Hospital, Ghent (Other)
Collaborators: MEDA Pharma GmbH & Co. KG (Industry); University of Wuerzburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-002865-40
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Bioavailability Study
Keywords: MP29-02
MeSH Terms: interventions — MP29-02; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational product (Experimental): MP29-02 137
  Interventions: Drug: MP29-02
- Non-investigational product (Active Comparator): fluticasone propionate
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: MP29-02 — local nasal application
  Other Names: Dymista
  Arms: Investigational product
Drug: Fluticasone propionate — local nasal application
  Other Names: FP
  Arms: Non-investigational product

SUMMARY:
The aim of this study is to investigate and to compare the bioavailability of MP29-02 and fluticasone propionate in nasal tissue after nasal application. This may provide a rational basis for the use of 1 puff per nostril dosage regimen of the drugs. Clinical experience has demonstrated the efficacy of the twice-daily treatment; however, so far, no data are available on the local tissue concentrations of MP29-02 after topical application.

DETAILED DESCRIPTION:
The study will be a single-centre, two-treatment half-side comparative open-label trial; all subjects will receive Dymista® or Flixonase Aqua in one nostril each.

Nasal tissue samples will be obtained from 24 patients. Subjects will be selected based on the subjects plan to undergo septoplasty, septorhinoplasty, or functional endoscopic sinus surgery. Subjects with different diagnoses can be added in the study: non-allergic rhinitis, allergic rhinits, chronic sinusitis and nasal polyposis. The number of subjects is based on a previous experiment where the presence of fluticasone propionate was tested on human nasal mucosal surface and in human nasal tissue after nasal application (Bonsmann, 2001).

ELIGIBILITY:
Inclusion Criteria:

* - Male and female patients
* Age: 18 - 70 years (included)
* Subjects who need to undergo septoplasty, septorhinoplasty or functional endoscopic sinus surgery unrelated to this study
* Willing and able to provide informed consent

Exclusion Criteria:

* - Patients who are member of the staff or relatives thereof directly involved in the conduct of the protocol
* Participant in any other trial during the last 30 days
* Previous treatment with Dymista or any other topical corticosteroid spray or drops within the last month before the operation
* Previous treatment with systemic corticosteroid in the last 2 months before operation
* Previous treatment with anti-histaminics 7 days before operation
* Pregnant or breast feeding women
* Allergic for one of the compounds azelastinehydrochloride or fluticasonpropionate
* Significant co-morbidity (for instance, but not limited to):

  * Glaucoma, cataracts, and increased intraocular pressure.
  * Subjects with active or quiescent tuberculosis; fungal, bacterial, viral, or parasitic infections; or ocular herpes simplex
  * Subjects with severe liver disease
* Use of prohibited concomitant medication

  * Potent inhibitors of cytochrome P450 (CYP) 3A4
  * Ritonavir
* Patients unwilling or unable to attend the proposed visit schedule
* Patients suspected or known not to be trustworthy or who are likely not to comply with the study directives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
bioavailability of MP29-02 in human nasal mucosa compared to commercially available fluticasone propionate | 1 hour
  bioavailability of both medicines will be tested in nasal mucosa and nasal secretion 1 after application

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, Principal Investigator — Upper Airways Research Laboratory, Department of Oto-Rhino-Laryngology, Ghent University Hospital, Ghent, Belgium.
Locations (1):
- University Hospital Ghent, departement otorhinolaryngology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No